CLINICAL TRIAL: NCT00121654
Title: Randomized Study on SCS for the Treatment of Refractory Angina Pectoris
Brief Title: Spinal Cord Stimulation (SCS) in Refractory Angina
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Gaetano Antonio Lanza, Università Cattolica del Sacro Cuore, Roma
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ITA-SCS1
Record Dates: First submitted 2005-07-14; First posted 2005-07-21 (Estimated); Last update posted 2009-03-10 (Estimated); Status verified 2009-03

CONDITIONS: Angina Pectoris
Keywords: Angina pectoris; Spinal cord stimulation; Refractory angina pectoris
MeSH Terms: conditions — Angina Pectoris | interventions — Spinal Cord Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): paresthesic SCS
  Interventions: Device: Spinal cord stimulation
- 2 (Active Comparator): subliminal SCS (75-80% of paresthesic threshold)
  Interventions: Device: Spinal cord stimulation
- 3 (Sham Comparator): low stimulation, consisting of an hour of SCS a day at 0.05 mV intensity, which does not have any significant stimulator effect (sham stimulation)
  Interventions: Device: Spinal cord stimulation

INTERVENTIONS:
Device: Spinal cord stimulation — Under sterile conditions and local anesthesia, the epidural space is punctured at the level of T5-T6 and a quadripolar electrode catheter is introduced and advanced under X-ray control into the epidural space. A suitable position for the electrode catheter is sought for, corresponding to the site where a prickling sensation (paresthesia) is felt and covers the area of radiation of angina pain under neurostimulation. The electrode catheter is connected to an internal pulse generator placed in a subcutaneous abdominal or gluteal pocket through an extension lead connected to the electrode by subcutaneous tunneling.

SUMMARY:
The study aims at assessing safety and efficacy of Spinal Cord Stimulation (SCS) for the treatment of refractory angina pectoris in a single blind, prospective, multicenter study.

Sixty patients with refractory angina with new SCS device implantation will be randomized to one of three treatment groups:

* paresthesic SCS;
* subliminal SCS;
* low (non effective) stimulation (control).

Clinical follow-up will be done at 1 and 3 months. Control group patients will then be randomized to paresthesic SCS or subliminal SCS for another 3 months and the 2 groups will be reassessed at 6 months.

DETAILED DESCRIPTION:
Aim of the study is to assess safety and efficacy of Spinal Cord Stimulation (SCS) for the treatment of refractory angina pectoris in a single blind, prospective, multicenter study. The study also assesses whether subliminal SCS may be as effective as paresthesic SCS in these patients.

Sixty consecutive patients with refractory angina with a new SCS device implantation will be randomized to one of three treatment groups:

* paresthesic SCS (group 1);
* subliminal SCS (75-80% of paresthesic threshold; group 2);
* low stimulation, consisting of an hour of SCS a day at 0.05 mV intensity, which does not have any significant stimulator effect (sham stimulation, group 3).

Study Procedure

Medical history, clinical data, drug therapy, Angina Canadian Cardiovascular Society (CCS) classification, Seattle Angina Questionnaire (SAQ), quality of life estimation by EuroQoL scale, detailed evaluation of angina attacks (frequency, intensity, duration of episodes; nitrates assumption) according to a structured diary, number of hospitalizations, emergency room (ER) admissions and cardiological visits in the previous 6 months and treadmill exercise stress test results will be obtained at the baseline visit.

Patients fulfilling inclusion criteria will undergo SCS implant. During the implant, stimulation tests will be performed to check paresthesic coverage of angina pain chest area.

Patients with adequate paresthesias will be randomized to one of the 3 groups. Follow-up visits will be performed at 1, 3, 6, and 12 months after the SCS implant. Drug therapy will not be changed at least during the first 3 months.

Patients assigned to group 2 (subliminal SCS) and those assigned to group 3 (sham SCS) will be blinded about the assigned treatment.

After the 3 months group 3, patients will be randomized to group 1 or group 2 and reassessed at 6-month follow-up (comparison between paresthesic versus subliminal SCS).

The controlled study will end at the 6-month follow-up, when each investigator will decide for the best stimulation for individual patients. Every patient will then be followed until 12 months from SCS implant.

Clinical assessment will be done at each follow-up visit. Exercise stress test results will be repeated at 3-, 6- and 12-month follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Stable angina pectoris refractory to optimal medical therapy, with at least 10 angina episodes in the three weeks previous SCS implant;
* Documentation of coronary artery disease and reversible myocardial ischaemia;
* Patient is not a candidate for or refuses surgical or percutaneous coronary revascularization;
* Availability for follow-up visits;
* Written informed consent.

Exclusion Criteria:

* Severe spinal cord diseases that prevent the catheter positioning in the epidural space;
* No paresthesic coverage of angina pain area during SCS;
* Unstable angina pectoris;
* Female patients in fertile age;
* Enrolment in other studies;
* Need for anticoagulant therapy;
* Patients needing diathermy treatment;
* Life expectancy <12 months.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2005-07; Primary Completion 2008-12 (Actual); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Reduction of angina symptoms | 1, 3, 6 and 12 months
improvement of quality of life | 1, 3, 6 and 12 months

SECONDARY OUTCOMES:
Improvement of exercise induced myocardial ischemia | 3, 6 and 12 months
evaluation of adverse events and complications | 0, 1, 3, 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano A Lanza, MD, Principal Investigator — Catholic University of the Sacred Heart
Locations (1):
- Istituto di Cardiologia - Università Cattolica del Sacro Cuore, Roma, Italy